CLINICAL TRIAL: NCT04710173
Title: Establishment of a Early Risk Model of Extracorporeal Membrane Oxygenation（ECMO） in Children With Acute Respiratory Distress Syndrome （ARDS） in China
Brief Title: Establishment of a Early Risk Model of ECMO in Children With ARDS
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Collaborators: The Children's Hospital of Zhejiang University School of Medicine (Other); Children's Hospital of Chongqing Medical University (Other); Guangdong Provincial People's Hospital (Other); Chinese PLA General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: fdpicu-07
Record Dates: First submitted 2021-01-12; First posted 2021-01-14 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: ARDS
Keywords: ECMO; ARDS; pediatric

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 2 ml whole blood in EDTA tube
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ARDS children: children with severe ARDS
  Interventions: Procedure: ECMO

INTERVENTIONS:
Procedure: ECMO — VV-ECMO

SUMMARY:
The key problem in the treatment of ARDS is refractory hypoxemia. Extracorporeal Membrane Oxygenation (ECMO) is an extracorporeal oxygenation of venous blood to eliminate carbon dioxide and return to the body. It has been an important part of the rescue treatment for ARDS. This study intends to explore the timing of ECMO. The main research hypothesis is that the appropriate timing of ECMO treatment can improve the weaning success rate and survival rate of children with severe ARDS; it is expected to provide a basis for determining the best timing of ECMO treatment

DETAILED DESCRIPTION:
Severe acute respiratory distress syndrome (ARDS), especially those caused by severe viral pneumonia, is still an important factor in the death of children, with a case fatality rate of 55%. The treatment includes lung protective ventilation and advanced ventilation support, but the effect is still not ideal for severe patients. ECMO can effectively support the respiratory system and provide good oxygen exchange. However, the survival rate of ECMO treatment in children with ARDS has a large bias.One of the key factors is the uneven timing of ECMO activation, which significantly affects the prognosis.This study intends to design a multi-center, prospective, non-randomized controlled trial , through retrospective research to find relevant factors affecting the prognosis of ECMO treatment, and to screen key indicators related to the timing of intervention; through a prospective cohort study to screen Good indicators and cut-off values suitable for starting ECMO , constructing and verifying comprehensive prediction models.

ELIGIBILITY:
Inclusion Criteria:

* Acute onset; within 7 days of clinical insult
* Chest imaging (radiograph or computed tomography) findings of new infiltrates (unilateral or bilateral) consistent with acute parenchymal disease
* Edema not fully explained by fluid overload or cardiac failure
* May present as new acute lung disease in setting of chronic lung disease and/or heart disease
* OI≥16
* Viral etiology is clear

Exclusion Criteria:

* Perinatal lung disease
* Large intracranial bleed with mass effect or need for neurosurgical intervention
* Hypoxic cardiac arrest without adequate CPR
* Irreversible underlying cardiac or lung pathology (and not a transplant candidate)
* Pulmonary hypertension and chronic lung disease
* Chronic multiorgan dysfunction
* Incurable malignancy
* Allogenic bone marrow recipients with pulmonary infiltrates
* Hepatic or renal failure
* Pertussis infection in infants
* Fungal pneumonia
* Immunodeficiency

Ages: 28 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children with acute respiratory distress syndrome（ARDS） admitted to the pediatric intensive care unit（PICU） of all the study centers
Sampling Method: Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Survival rate | 28 days after hospital discharge
  The survival rate of children in 28 days after hospital discharge

SECONDARY OUTCOMES:
ECMO weaning rate | 48 hours after ECMO weaning
  The success of ECMO weaning is defined as the survival of patients after ECMO weaning for 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ye Cheng, doctor, Study Director — Children's Hospital of Fudan University
Locations (3):
- China (3):
  - Chinese PLA General Hospital, Beijing
  - Children's Hospital of Chongqing Medical University, Chongqing
  - Guangdong Provincial People's Hospital, Guanzhou